CLINICAL TRIAL: NCT00186212
Title: Alternative Support for Rural and Isolated Women in an HMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Cheryl Koopman, Ph.D., Professor (Research), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5BB-1801
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Stress Disorders, Post-traumatic; Depression; Breast Cancer
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: workbook/journal on coping with breast cancer
Behavioral: standard educational materials on breast cancer

SUMMARY:
Evaluate the effects of a workbook/journal for helping isolated women to cope with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) is a woman; and 2) has been diagnosed with primary breast cancer

Exclusion Criteria:

* 1) is under 18; or 2) can not speak and read in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-09; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
depression
posttraumatic stress disorder

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Koopman, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States